CLINICAL TRIAL: NCT02041117
Title: Resuvastatin Treatment for Symptomatic Middle Cerebral Artery Stenosis Based on High-resolution Magnetic Resonance Imaging in Two Years
Brief Title: Resuvastatin Treatment for Symptomatic Middle Cerebral Artery Stenosis Based on High-resolution Magnetic Resonance Imaging
Acronym: REALM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Executive Vice-President, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012ZX09303-005-001
Record Dates: First submitted 2014-01-02; First posted 2014-01-20 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Intracranial Arterial Stenosis
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosuvastatin (Other)
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin, 10mg for 4-weeks, then according to the results of the LDL-C, adjust dose of rosuvastatin, maximum to 20 mg/d, to reduce LDL-C under 70 mg/dl for two years.
  Other Names: Crestor

SUMMARY:
1. It is a multicenter, open-label, sing arm study to evaluate the effects of treatment of Rosuvastatin 10-20mg in volume and morphology of atherosclerotic plague by reducing LDL-C level to or less than 70mg/dl.
2. Ischemic stroke patients will be enrolled within 1 month after stroke onset.
3. Patients will be visited at 0m, 1m, 3m, 6m, 9m, 12m, 18m and 24m.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 18 and 75 years of age.
2. Ischemic stroke originate from middle cerebral artery(MCA) AS stenosis, stroke onset within 1 month.
3. LDL-C level is more than 70mg/dl (1.8mmol/L), but less than 250mg/dl (6.5mmol/L); and triglyceride level is less than 353mg/dl (4.0mmol/L).
4. total term of statin therapy less than 2 month in past 1year before entering the study.

（5）30-70% intracranial artery stenosis in M1 segment of MCA comfirmed by CTA or MRI at least 1 or more atherosclerotic plaques in M1 segment of MCA is detectable.

（6）Female patients must agree to use an effective form of birth control throughout the 2-year study treatment period.

（7）The patients who are willing to be enrolled have to remain on the low cholesterol dietary for the study duration.

（8）The patient must be able to comply with scheduled visits, the treatment plan and all laboratory tests.

（9）Written informed consent is provided to participate in the study.

Exclusion Criteria:

1. Any hemorrhagic stroke or hemorrhagic infarction
2. Presence of any of cardiac sources of embolism
3. Ischemic stroke caused by non MCA stenosis
4. The patients has LDL cholesterol ≤ 70mg/dl or familial hypercholesterolemia.
5. Previous treatment of target lesion with a stent, angioplasty, or other mechanical device, or plan to perform staged angioplasty within 2 years
6. Any aneurysm proximal to or distal to stenotic intracranial artery
7. Intracranial tumor (except meningioma) or any intracranial vascular malformation
8. Thrombolytic therapy within 24 hours before enrollmentnt
9. The patient has plans for surgical/endovascular intervention for intracranial, carotid, coronary and/or peripheral arterial disease during the course of the study.
10. The patient has or is being treated or evaluated for diagnosed tuberculosis.
11. The patient has a history of malignant neoplasm within the previous 5 years (exception: curable non-melanoma skin malignancies).
12. The patient has a known immunodeficient state (e.g., human immunodeficiency virus) or is being treated with immunosuppressive drugs including cyclosporine.
13. The patient has any other clinically significant medical condition that, in the opinion of the Investigator, could impact the patient's ability to successfully complete the trial.
14. Life expectancy of patients is less than 2 years.
15. The patient have to take medicines as follow: Hormonal therapy, Cyclosporine and other lipid lowering agents: fish oil, garlic essential oil etc.
16. The patient has a history of recent alcohol abuse, drug abuse or significant mental illness.
17. The patient has any condition that would prevent the patient from giving voluntary informed consent.
18. The patient has an inability to tolerate oral medication administration.
19. The patient has a known or suspected allergy to the study medication(s) or the class of study medication to be administered.
20. The patients cannot finish HR-MRI for any reasons.
21. Pregnancy or of childbearing potential and unwilling to use contraception for the duration of this study
22. The patient is enrolled or plans to enroll in another clinical drug or device/interventional trial during this study.
23. The patient has the history of epilepsy/seizures.
24. The patient has liver function tests > 1.5 times the upper limit of normal, serum creatinine > 2.0 mg/dL, GFR < 30 ml/min or has abnormal laboratory values which are deemed clinically significant by the investigator.
25. The patient has the history of myopathy.
26. The patient has thyroid stimulating hormone > 1.5xULN.
27. BMI ≥ 30 kg/m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2014-02-24 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
The change in the percentage of volume of MCA atherosclerosis plaque after 2 years treatment of Rosuvastatin 10-20mg | 2 year

SECONDARY OUTCOMES:
The change in Percentage of plaque volume of M1segment plaque | 6 months and 1 year
The change in Percentage of lumen volume | 2 years
The change in percentage of lipid rich necrotic core | 2 years
Recurrency of stroke or TIA | 2 years
The change of percentage in LDL-C from baseline | 2 years
The change in HDL-C level from baseline | 2 years
To explore the relationship between the change of plaque volumn and morphology and the change in LDL-C, HDL-C and Hs-CRP level | 2 years
safety-Rhabdomyolysis，Hepatonecrosis | 2 years
The change in percentage of thickness of fibrous cap | 2 years
The change in percentage of intraplaque hemorrhage | 2 years
The change in hsCRP level from baseline | 2 years
2.Severe bleeding incidence (GUSTO definition), including fatal bleeding and symptomatic intracranial hemorrhage | 2 years
Incidence symptomatic and asymptomatic intracranial hemorrhagic events at 3 months | 2 years
Moderate bleeding (GUSTO definition) | 2 years
Intracranial hemorrhage | 2 years
Total mortality | 2 years
AEs/SAEs reported by the investigators | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital affliated to Capital Medical University, Beijing, Beijing Municipality, China